CLINICAL TRIAL: NCT02791126
Title: Curvedness-based Imaging: A Novel Automated & Comprehensive Approach for Ventricular Function Assessment in Heart Failure
Brief Title: A Novel Automated & Comprehensive Approach for Ventricular Function Assessment in Heart Failure
Status: Completed | Type: Observational
Sponsor: National Heart Centre Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: 2013/934/C
Record Dates: First submitted 2016-05-31; First posted 2016-06-06 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2017-09

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Heart Failure: Patients presented to hospital with a primary diagnosis of Heart Failure or are attending a hospital clinic for management of Heart Failure within 6 months of an episode of decompensated heart failure, which either resulted in a hospital admission (primary diagnosis) or was treated in out-patient clinic.
  Cardiovascular Magnetic Resonance and Echocardiogram will be performed.
  Interventions: Other: Cardiovascular Magnetic Resonance; Other: Echocardiogram

INTERVENTIONS:
Other: Cardiovascular Magnetic Resonance — For the evaluation of left ventricular volumes, function and mass. This is also for the assessment of myocardial fibrosis based on delayed enhancement imaging technique.
Other: Echocardiogram — For the assessment of diastolic and systolic function as well as valvular and cardiac function. Ventricular-arterial coupling will also be performed.

SUMMARY:
Heart failure is a major health care burden. It can occur with either normal or reduced LV ejection fraction, depending on different degrees of ventricular remodelling. The investigators recently published a new method, curvedness-based imaging. The investigators have also reported the diagnostic utility of curvedness-based imaging in various cardiac diseases. The investigators now propose to prospectively assess curvedness-based imaging for diagnosis of heart failure with normal ejection fraction and with reduced ejection fraction, and examine left ventricular systolic and diastolic function and predicts the prognosis in a cohort of HF patients.

DETAILED DESCRIPTION:
Heart failure imposes major global health care burden on society and suffering for the individual.In the US, HF affects 5.7 million patients, and is the leading cause of hospitalization for people over 65 years, with 25% to 50% rate or hospital readmission within 6 months.In Singapore, between 1991 and 1998, it accounted for 4.5% of all hospital admissions and 2.5% of mortality in the geriatric age group.It confers an annual mortality of 10%.

The early diagnosis and identification of the underlying etiology of HF is of paramount importance; some causes require specific treatment and may be correctable. From updated American College of Cardiology/American Heart Association guidelines, some questions must be addressed for suspected HF patients: Is the left ventricular ejection fraction preserved or reduced? Is the structure of the LV normal or abnormal? Are there other structural abnormalities such as right ventricular (RV) abnormalities that could account for the clinical presentation? Is there LV global and regional dysfunction and to what extent? Is the etiology ischemic or non-ischemic?

Cardiac imaging is important both for HF diagnosis and monitoring of progress. Impaired pump function, expressed reduced left ventricular ejection fraction is often used as a marker of HF. About 50% of HF have preserved EF.In this situation, more intricate and comprehensive imaging involving measurement of multiple diastolic and systolic parameters, usually using echocardiography, may become necessary to address the questions mentioned above.

Our solution is expected to result in a significant cost saving for HF patients. HF diagnosis is still very challenging, consisting of assessment of medical and family histories, a physical exam and diagnostic imaging tests. The investigators compare the cost difference in traditional way against our proposed solution. The traditional diagnostic tests include chest x-ray, BNP blood test, echocardiography, nuclear heart scan and cardiac catheterization. In this project, the investigators estimate the cost of echocardiography, nuclear heart scan and cardiac catheterization for HF diagnosis. Based on clinical experience, among 1000 patients undergoing echocardiography, 50% will be referred to nuclear heart scan and 30% will be referred to invasive cardiac catheterization. The cost of the whole workup is estimated to be $1.95 million. If 1000 patients undergo our proposed CBI solution directly, the cost estimated at $1.4 million. The cost saving is estimated at S$400 per patient.

Hence, the investigators will be exploring the following for this study:

Primary aim: Assess LV systolic and diastolic function from curvedness-based imaging in 120 HF patients with reduced ejection fraction and normal ejection fraction.

Secondary aim: Evaluate the utility of curvedness-based imaging for the diagnosis of etiology of HF, against gold standard gadolinium enhanced CMR in subgroup of HF patients.

Exploratory aim: Evaluate the utility of curvedness-based imaging for the prediction of prognosis during 6 month follow up, where clinical outcome include death, CV death and HF re-admission.

ELIGIBILITY:
Inclusion Criteria:

* Patients presented to hospital with a primary diagnosis of Heart Failure or are attending a hospital clinic for management of Heart Failure within 6 months of an episode of decompensated heart failure, which either resulted in a hospital admission (primary diagnosis) or was treated in out-patient clinic.
* Written informed consent obtained

Exclusion Criteria:

* Aged < 21 years
* Contraindication to CMR examination.
* Cardiac pacemaker
* Brain aneurysm or clips
* Electronic implants or prosthesis
* Eye metal foreign body injury
* Severe claustrophobia
* Severe renal impairment, glomerular filtration rate < 30ml/min/1.73m2
* Non-cardiac illness with life expectancy of less than 2 years
* Previous heart, kidney, liver or lung transplantation.
* HF primary due to severe valve disease
* Other specific subgroups of HF: Including constrictive pericarditis, complex adult congenital heart disease, hypertrophic cardiomyopathy, eosinophilic myocarditis, cardiac amyloid and acute chemotherapy-induced cardiomyopathy.
* Isolated right heart failure. Combined right and left heart failure will be included; Secondary to severe lung disease or pulmonary hypertension.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presented to hospital with a primary diagnosis of Heart Failure or are attending a hospital clinic for management of Heart Failure within 6 months of an episode of decompensated heart failure, which either resulted in a hospital admission (primary diagnosis) or was treated in out-patient clinic
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2013-11; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Allergic reaction due to MRI contrast | Within first day of scan

CONTACTS AND LOCATIONS:
Overall Officials: Ru San Tan, MD, Principal Investigator — National Heart Centre Singapore
Locations (1):
- National Heart Centre Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No